CLINICAL TRIAL: NCT05670977
Title: A Randomized, Double Blind, Controlled Study of Improved Skin Anti-aging Outcomes Associated With Collagen Fortified Consumption In 30 to 50-Year-old Women
Brief Title: Improved Skin Anti-aging Outcomes Associated With Collagen Fortified Consumption In 30 to 50-Year-old Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong HuaPeptides Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-SM-12-HT-001
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Skin Laxity; Skin Lines
Keywords: Collagen; skin anti-aging; skin moisture; skin elasticity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study product plus collagen supplement (Active Comparator): 5g/bag, containing the following ingredients per 5g serving:
  * Collagen tripeptide 1500 mg
  * Elastin peptide 150 mg
  Interventions: Dietary Supplement: Study product plus collagen supplement
- Study product without collagen supplement (Placebo Comparator): 5g/bag, containing the following ingredients per 5g serving:
  * Peach juice 8 mg
  * Erythritol 10 mg
  Interventions: Dietary Supplement: Study product without collagen supplement

INTERVENTIONS:
Dietary Supplement: Study product plus collagen supplement — The participants in this arm will use the assigned product for 2 months, 5g one time, once a day.
  Arms: Study product plus collagen supplement
Dietary Supplement: Study product without collagen supplement — The participants in this arm will use the assigned product for 2 months, 5g one time, once a day.
  Arms: Study product without collagen supplement

SUMMARY:
The goal of this clinical trial is to study the efficacy of collagen supplement on the moisture content and elasticity.

70 participants of 30-50 years old women will be enrolled from two study sites and randomly assigned to use two products (study product plus collagen supplement and placebo product without collagen supplement) for 2 months.

Researchers will compare the two groups to validate the assumption that there is significant improvement on skin anti-aging effect for participants using study product plus collagen supplement.

DETAILED DESCRIPTION:
This study is two arms, randomized, double-blind controlled trial. There will be two study sites and 35 eligible participants at each study site will be enrolled with the expectation of having 30 participants completed per study group. Particants will be randomly allocated to use one of the two study products defined in the trial protocol for two months. Up to three study visits will be made by the participant over a 2-month period. All relevant data will be captured and recorded into CTMS (Clinical Trial Management System). The data will be analyzed and reported after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Chinese females, age between 30-50;
* Be in general good health;
* Understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate;
* Have mild to moderate darker skin tone 3 on Unilever visual scale of 1~9;
* Have mild pigmentation level 2 on Unilever visual scale of 0~9;
* Have visual grading score on crow's feet 3 on Unilever visual scale of 0~9;
* Have visual grading score on peri-oral 3 on Unilever visual scale of 0~9;
* Have visual grading score on nasolabial folds 3 on Unilever visual scale of 0~9;
* Tolerate to well-known anti-aging actives;
* Agree to not use any other creams, lotions, moisturizers on the face, other than what is provided for the duration of the study;
* Agree to refrain from wearing make-up (such as foundation, eye shadow, lipstick etc.) or any skin care products on the face on the study visits;
* Agree to avoid washing the treatment site area for two hours following product application and agree to avoid washing appliances (i.e., sponge, wash cloth, loofah, etc.).

Exclusion Criteria:

* Have used any skin lightening /anti-aging benefits products at least one month before this study
* Subject having done facial injections and/or aesthetic surgery.
* Be involved in any aspect of test administration, i.e., evaluating or overseeing activities related to product.
* Have participated in any clinical study involving the test sites within the previous 6 months, or is subject participating in any clinical study concurrently.
* Have a history of any type of bagcer, including but not limited to any type of skin bagcer (squamous or basal cell carcinoma at the treatment site) or history of malignant melanoma at any body site.
* Have a history of skin disease or the presence of a skin condition on the test sites that the Investigator feels would interfere with the study.
* Be taking antihistamines (> 3x/week) or anti-inflammatory (> 8x/week) on a regular basis, or has the subject taken systemic or topical steroidal medications within 4 weeks of study enrolment.
* Have any of the following conditions or factors that the investigator believes may affect the response of the skin or the interpretation of the test results, including, but not limited to, diabetes, pregnancy, lactation.
* Have any cuts/abrasions on the test site at baseline.
* Have had a suspicious skin lesion removed by a dermatologist at any time.
* The subject is an employee of sponsor or the site conducting the study.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be women of 30-50 years old
Enrollment: 70 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Skin Elasticity | baseline day 0, day 60
  The changes of skin elasticity from baseline to day 60 by CK Cutometer MPA580
Skin Moisture | baseline day 0, day 60
  The changes of skin moisture from baseline to day 60 by Corneometer CM 825

SECONDARY OUTCOMES:
Skin Barrier | baseline day 0, day 30, day 60
  The changes of skin barrier in terms of TEWL (Trans Epidermal Water Loss) by Aquaflux F200
Lines/Wrinkles | baseline day 0, day 30, day 60
  The changes of the lines/wrinkles on the face by Miravex Antera 3D imaging system
Facial Glow | baseline day 0, day 30, day 60
  The changes of Facial Glow by expert visual assessment
Skin Diagnosis | baseline day 0, day 30, day 60
  The skin diagnosis (4 modes and 2 side views) with VISIA CR Facial Imaging System

CONTACTS AND LOCATIONS:
Overall Officials: Yun Wang, MD, Principal Investigator — NO. 9 Hospital affiliated to Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Ai'er Hospital, Shanghai, Shanghai Municipality
  - SPRIM Central Lab, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proksch E, Segger D, Degwert J, Schunck M, Zague V, Oesser S. Oral supplementation of specific collagen peptides has beneficial effects on human skin physiology: a double-blind, placebo-controlled study. Skin Pharmacol Physiol. 2014;27(1):47-55. doi: 10.1159/000351376. Epub 2013 Aug 14. PMID 23949208
- [Background] Proksch E, Schunck M, Zague V, Segger D, Degwert J, Oesser S. Oral intake of specific bioactive collagen peptides reduces skin wrinkles and increases dermal matrix synthesis. Skin Pharmacol Physiol. 2014;27(3):113-9. doi: 10.1159/000355523. Epub 2013 Dec 24. PMID 24401291
- [Background] Shariff R, Du Y, Dutta M, Kumar S 5th, Thimmaiah S, Doraiswamy C, Kumari A, Kale V, Nair N, Zhang S, Joshi M, Santhanam U, Qiang Q, Damodaran A. Superior even skin tone and anti-ageing benefit of a combination of 4-hexylresorcinol and niacinamide. Int J Cosmet Sci. 2022 Feb;44(1):103-117. doi: 10.1111/ics.12759. Epub 2022 Feb 1. PMID 34958693
- [Background] Wang L, Xu YN, Chu CC, Jing Z, Chen Y, Zhang J, Pu M, Mi T, Du Y, Liang Z, Doraiswamy C, Zeng T, Wu J, Chen L. Facial Skin Microbiota-Mediated Host Response to Pollution Stress Revealed by Microbiome Networks of Individual. mSystems. 2021 Aug 31;6(4):e0031921. doi: 10.1128/mSystems.00319-21. Epub 2021 Jul 27. PMID 34313461
- [Background] Du Y, Doraiswamy C, Mao J, Zhang Q, Liang Y, Du Z, Vasantharaghavan R, Joshi MK. Facial skin characteristics and concerns in Indonesia: A cross-sectional observational study. Skin Res Technol. 2022 Sep;28(5):719-728. doi: 10.1111/srt.13189. Epub 2022 Jul 4. PMID 35785442